CLINICAL TRIAL: NCT06276192
Title: Digital Physiotherapy Treatment for Patients With Subacromial Pain Compared to Traditional Physiotherapy Treatment in Primary Care - a Non-Inferiority Randomised Controlled Trial
Brief Title: Digital Physiotherapy Treatment for Patients With Subacromial Pain Compared to Usual Physiotherapy in Primary Care
Acronym: diSAID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Teresa Holmgren, PhD Physical therapist, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-01882-01
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Subacromial Pain Syndrome; Shoulder Pain; Rotator Cuff Syndrome
Keywords: Shoulder pain; Subacromial pain; Digital care; Digital health intervention; Physiotherapy; Primary care
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Non-Inferiority Randomised Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Physiotherapy (diSAID) (Experimental): The digital physiotherapy group receives the digital Shoulder Aid (diSAID) strategy available via a web application. For three months, this group will complete a home-based rehabilitation programme containing education and evidence based exercises for patients with subacromial pain tutored by videos, images and instructions.The treatment is standardized but can be customized by a responsible physiotherapist during the whole treatment period. The Physiotherapist also deliver progression in the education and in the exercises during the whole treatment period and can support the patient via a messenger function in the web application.
  Interventions: Other: Digital Physiotherapy (diSAID)
- Traditional Physiotherapy (Active Comparator): The traditional physiotherapy group receives current practice provided by physiotherapist in primary care with no predefined directives. The treating physiotherapist are instructed to treat their patient as they usually do.
  Interventions: Other: Traditional Physiotherapy

INTERVENTIONS:
Other: Digital Physiotherapy (diSAID) — The diSAID is developed by the research group and is a modified version of a previously tested exercise program for patients with subacromial pain. The diSAID is distributed in three stages with; Information about subacromial pain, effects of exercise, pain management and ergonomics in everyday living and at work. The training includes exercises for the rotator cuff and scapular stabilizers as well as posterior shoulder stretch. The exercises are performed 1 time/day during twelve weeks with a progression of dose, load and complexity continuously. Pain while performing the exercise program is accepted up until NRS 5 out of 10.
  During ongoing treatment, there is the opportunity for counselling, individualization of exercises, adjustment of dose and load based on stated instructions from the treating physiotherapist.
  Adherence, levels of pain and function is reported continuously by the patient via the digital platform.
  Arms: Digital Physiotherapy (diSAID)
Other: Traditional Physiotherapy — Patients in the active control group are offered the usual treatment practice that is currently offered by physiotherapists in primary care. No predetermined directives for the active control group are defined prior to the study and can contain; home exercise programs, manual therapy and other techniques. The treating physiotherapists in this group are not involved in the digital treatment. The choice of interventions, amounts of visits and adherence is checked retrospectively via patient data and medical records.
  Arms: Traditional Physiotherapy

SUMMARY:
The goal of this clinical trial is to test a digital treatment for patients with subacromial pain using the digital Shoulder Aid (diSAID) strategy. The participants in this study will be randomly assigned to digital treatment (diSAID) or to receive the treatment that is currently available in primary care, i.e. continue according to usual practice.

The main question this clinical trial aims to answer are:

- Can the diSAID improve shoulder function and reduce pain for patients with subacromial pain in primary care?

DETAILED DESCRIPTION:
Subacromial pain is the most common shoulder complaints in the general population. The pathology is multifactorial and mainly explained by pain generated from structures in the space between the caput humeri and acromion, especially the bursa and tendons of the rotator cuff. Exercises have positive effects on shoulder function, pain and satisfaction in patients with subacromial pain and is according to current evidence the primary treatment for this condition. Surgery and exercise have been shown to have an equivalent positive effect and it is possible to avoid surgery with specific training. This means that the motive for surgery has become increasingly questionable. Despite this, many patients undergo surgery without having taken part in specific supervised training and the selection of patient's prior to surgery is still inadequate. One reason for this may be that resources in healthcare are limited. Supervised training with physical visits over a longer period of time can be difficult for the primary care to offer. This require demands on physiotherapists' skills, time and resources.

Clinical studies with digital solutions are increasing and occur in several areas of healthcare. Digital interventions have proven to be effective in several diseases and disorders and can increase access to health education in a cost-effective way.

This is a single-blind, prospective, non-inferiority randomised controlled trial, designed to evaluate the feasibility and efficacy of a digital physiotherapy treatment compared to traditional physiotherapy for patients with subacromial pain in a primary care setting. The hypothesis is that clinical outcomes of the digital physiotherapy intervention for patients with subacromial pain can be effective and non-inferior compared to traditional physiotherapy in primary care.

Further the study objective is to evaluate the cost-effectiveness and impact on the environment using a digital intervention.

Sample size calculation: The estimated sample size is based the primary outcome SPADI assuming α = 0.05, β = 0.2 with a given power of 80% and a standard deviation of 18. A non-inferiority margin is set to 10 points (δ = -10) in total SPADI scores. Consequently, 82 patients have to be included, 41 per treatment group. Due to drop outs an over recruitment is planned (Total achievement of 60 per group).

We will use unpaired t-tests to compare the effect of treatment between the different groups regarding the primary outcome shoulder function and pain evaluated with SPADI after 3 months. The H0 hypothesis will be rejected and the H1 hypothesis will be accepted if a significant difference is proven. H0 is also rejected if non-inferiority of digital physiotherapy to traditional physiotherapy is proven. This is declared when the upper confidence limit of the one-sided confidence interval for the mean change of SPADI is lower than the selected non-inferiority margin (δ = -10).

(H0 : μA - μB ≤ -δ; H1 : μA - μB ≥ -δ).

Method:

Patients with subacromial pain are recruited from five different physiotherapy units in county of Region Östergötland, in Sweden. All patients receives an in-person evaluation performed by physiotherapists in primary care to ensure that potential participants meet the eligibility criteria. Participants available for recruitment due to study criteria's are assigned randomly to 1) Digital physiotherapy group 2) Traditional physiotherapy group. All participants will be followed-up after three months, six months and two years after the received intervention.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Pain duration >2 weeks
* Lateral shoulder pain (C5 dermatome)

At least three positive tests as follows:

* Painful arc
* External rotation resistance test
* Jobe's test
* Neer's impingement sign
* Hawkin's-Kennedy's impingement test

Exclusion Criteria:

* Symptoms are related to a traumatic event in the last 6 months with suspected rotator cuff tear, dislocation or fracture.
* Clinical features of cervical radiculopathy
* Clinical features of Adhesive capsulitis
* The patient does not understand or can not read Swedish
* The patient has no access to BankID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-26 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
Mean change in shoulder function and pain after 12 weeks using The Shoulder Pain and Disability Index (SPADI) | Initial, 12 weeks, 6 months, 2 year
  The Shoulder Pain and Disability Index has good psychometric properties with good reliability and validity. It consists of two sub-areas, the first area includes five questions for the estimation of pain and the second area includes eight questions about the impact on activity-related function of the upper extremity. Grading of pain or functional limitation goes from 0-10 where 0 indicates "no pain or disability" and 10 indicate "maximum pain or disability". The sub-areas generate individual scales as well as a common total score that is given as a percentage. Minimal Clinically Important Difference is 8 to 13 points and Minimal Detectible Change is 18 points.

SECONDARY OUTCOMES:
Mean change in shoulder pain intensity at rest, arm activity and at night measured by numeric rating scale (NRS) | Initial, 12 weeks, 6 months, 2 year
  Pain level is rated between 0-10, where 0 corresponds to "no pain" and 10 corresponds to "worst pain imaginable".
Mean change in pain Self-Efficacy | Initial, 12 weeks, 6 months, 2 year
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire assessing peoples capabilities and the confidence in performing activities while ongoing pain. Each task have an answer that range from "not at all confident" to "completely confident" on a 7-point scale. The questions includes capacity of specific functional tasks and beliefs of handling function demands. Added scores from all items gives a total score, ranging from 0 to 60. Higher scores reflect stronger self-efficacy. The PSEQ have good psychometric properties of reliability, validity, and internal consistency
Mean change of self-reported rating of improvement | Initial, 12 weeks, 6 months, 2 year
  Patient Global Impression of Change (PGIC) is a self-report measure reflecting a patient's improvement and belief about the efficacy of treatment between two time points. In this version the patients rate their change as "Completely recovered" "Much improved" "Slightly improved" "Unchanged" or "Worse".
Mean change of health-related quality of life | Initial, 12 weeks, 6 months, 2 year
  EuroQol Instrument (EQ5D index and EQ VAS) is a self-reported measure capturing five dimensions of health-related quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The questions are validated and reliable for a broad spectra of medical conditions. The instrument can also be used as a measure in Estimation of health utility and quality-adjusted life years (QALYs) and is a part of the economic evaluation of the digital treatment.

OTHER OUTCOMES:
Patients treatment expectancies | Initial
  Stanford Expectations of Treatment Scale (SETS) is used to assess expectancy effects. Patients rate their expectations before treatment on a 7-point scale with two sub-categories: negative and positive treatment expectancies. The instrument can be used to improve statistical sensitivity for detecting treatment differences or to identify patients with poor treatment expectancies.
Patients self-reported rating of pain sensitivity | Initail
  2. The Pain Sensitivity Questionnaire (PSQ) is a 17-item questionnaire that assesses a patient's perception to different fictional physical stimuli that might be experienced in daily life. The patient rate their imagined pain intensity of each item on an 11-point scale with 0 meaning "not painful at all" and 10 meaning "worst pain imaginable." The PSQ is a reliable and valid measure and can be expressed in PSQ-total score or PSQ-minor score.
  The Pain Sensitivity Questionnaire (PSQ) is a 17-item questionnaire that assesses a patient's perception to different fictional physical stimuli that might be experienced in daily life. The patient rate their imagined pain intensity of each item on an 11-point scale with 0 meaning "not painful at all" and 10 meaning "worst pain imaginable." The PSQ is a reliable and valid measure and can be expressed in PSQ-total score or PSQ-minor score.
Costs and cost-effectiveness direct and indirect | 3 months and 2 year
  The economic evaluation will primary be based on the time and amounts of visits causing cost for the health sector during the treatment. An economic analysis of QALYS, reduced remittance to specialised care and surgery will be analysed in a longer perspective.
Impact on the environment | 2 year
  Evaluation will we based on emission of CO2 connected to the treatments. The climate impact will primary be linked to the direct emissions per passenger kilometers (ie emissions from the fuel used in transport to care visits)

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Petersson, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF
Time Frame: A statistical analysis plan will be available at Clinicaltrials.gov prior to the start of data analysis.

REFERENCES:
- [Background] Vandvik PO, Lahdeoja T, Ardern C, Buchbinder R, Moro J, Brox JI, Burgers J, Hao Q, Karjalainen T, van den Bekerom M, Noorduyn J, Lytvyn L, Siemieniuk RAC, Albin A, Shunjie SC, Fisch F, Proulx L, Guyatt G, Agoritsas T, Poolman RW. Subacromial decompression surgery for adults with shoulder pain: a clinical practice guideline. BMJ. 2019 Feb 6;364:l294. doi: 10.1136/bmj.l294. PMID 30728120
- [Background] Holmgren T, Hallgren HB, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. Br J Sports Med. 2014 Oct;48(19):1456-7. doi: 10.1136/bjsports-2014-e787rep. PMID 25213604
- [Background] Hallgren HC, Holmgren T, Oberg B, Johansson K, Adolfsson LE. A specific exercise strategy reduced the need for surgery in subacromial pain patients. Br J Sports Med. 2014 Oct;48(19):1431-6. doi: 10.1136/bjsports-2013-093233. Epub 2014 Jun 26. PMID 24970843
- [Background] Clausen MB, Merrild MB, Holm K, Pedersen MW, Andersen LL, Zebis MK, Jakobsen TL, Thorborg K. Less than half of patients in secondary care adheres to clinical guidelines for subacromial pain syndrome and have acceptable symptoms after treatment: A Danish nationwide cohort study of 3306 patients. Musculoskelet Sci Pract. 2021 Apr;52:102322. doi: 10.1016/j.msksp.2021.102322. Epub 2021 Jan 12. PMID 33485212